CLINICAL TRIAL: NCT00000776
Title: Dexamethasone in Cryptococcal Meningitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 202; 11178 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Dexamethasone; Drug Therapy, Combination; Fluconazole; Flucytosine; Acquired Immunodeficiency Syndrome; Amphotericin B; Brain Diseases
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome; Brain Diseases | interventions — Flucytosine; Fluconazole; Amphotericin B; Dexamethasone

INTERVENTIONS:
Drug: Flucytosine
Drug: Fluconazole
Drug: Amphotericin B
Drug: Dexamethasone

SUMMARY:
To evaluate the effect of corticosteroids on reducing elevated intracranial pressure in cryptococcal meningitis. To evaluate the safety of corticosteroids in patients with cryptococcal meningitis and intracranial hypertension.

In AIDS patients with cryptococcal meningitis, a correlation has been found between early death and elevated intracranial pressure. Since dexamethasone has been found to reduce intracranial pressure resulting from other forms of meningitis, it may be of benefit in AIDS patients with cryptococcal meningitis.

DETAILED DESCRIPTION:
In AIDS patients with cryptococcal meningitis, a correlation has been found between early death and elevated intracranial pressure. Since dexamethasone has been found to reduce intracranial pressure resulting from other forms of meningitis, it may be of benefit in AIDS patients with cryptococcal meningitis.

Patients are randomized to receive dexamethasone or placebo every 6 hours for 72 hours (days 1 through 3). Additionally, standard antifungal therapy with amphotericin B and flucytosine is given for 2 weeks, followed by fluconazole for 8 weeks. Lumbar punctures will be performed daily on days 1 through 3, on days 7 and 14, and at week 10.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine or systemic chemoprophylaxis for PCP.
* Preventive therapy for steroid-associated ulcers and any other therapies required to manage steroid toxicity (e.g., insulin).

Patients must have:

* Documented initial episode or relapse of acute cryptococcal meningitis. (NOTE: Patients must be untreated for this episode except for administration of a test dose of 1 g or less amphotericin B.)
* Acute cryptococcal meningitis with cerebrospinal fluid opening pressure >= 250 mm H2O prior to receipt of antifungal therapy for this episode.
* Documented HIV infection OR a diagnosis of AIDS based on a documented AIDS-defining opportunistic infection.
* Ability to begin therapy within 8 hours after the pre-entry lumbar puncture.
* Consent of parent or guardian if less than 18 years of age.

NOTE:

* Comatose patients eligible provided informed consent can be provided by guardian or next of kin.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Concurrent CNS disease such as another infection or neoplasm that would interfere with assessment of response.
* Prison incarceration.

Concurrent Medication:

Excluded:

* Acetazolamide, mannitol, urea preparations, and other corticosteroids during the first 72 hours of the study.
* Treatment or prophylaxis with other systemic antifungal agents at any time.
* Antiretroviral therapy during the first 72 hours of the study.

Prior Medication:

Excluded within 7 days prior to study entry:

* Corticosteroids, mannitol, urea preparations, acetazolamide, or more than 24 hours of phenytoin.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Jacobson, Study Chair
Locations (14):
- United States (13):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
- Univ of Puerto Rico, San Juan, Puerto Rico